CLINICAL TRIAL: NCT03598998
Title: A Phase 1/2 Study of Pembrolizumab Plus Pralatrexate for Treatment of Relapsed or Refractory Peripheral T-Cell Lymphomas
Brief Title: Pembrolizumab and Pralatrexate in Treating Patients With Relapsed or Refractory Peripheral T-Cell Lymphomas
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17501; NCI-2018-01420 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 17501 (Other: City of Hope Medical Center)
Record Dates: First submitted 2018-07-16; First posted 2018-07-26 (Actual); Results first posted 2024-08-27 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Anaplastic Large Cell Lymphoma; Nodal Peripheral T-Cell Lymphoma With TFH Phenotype; Recurrent Anaplastic Large Cell Lymphoma; Recurrent Angioimmunoblastic T-Cell Lymphoma; Recurrent Enteropathy-Associated T-Cell Lymphoma; Recurrent Follicular Lymphoma; Recurrent Hepatosplenic T-Cell Lymphoma; Recurrent Mature T- Cell and NK-Cell Non-Hodgkin Lymphoma; Recurrent Monomorphic Epitheliotropic Intestinal T-cell Lymphoma; Recurrent Mycosis Fungoides; Recurrent Peripheral T-Cell Lymphoma, Not Otherwise Specified; Refractory Anaplastic Large Cell Lymphoma; Refractory Angioimmunoblastic T-Cell Lymphoma; Refractory Enteropathy-Associated T-Cell Lymphoma; Refractory Follicular Lymphoma; Refractory Hepatosplenic T-Cell Lymphoma; Refractory Mature T-Cell and NK-Cell Non-Hodgkin Lymphoma; Refractory Mycosis Fungoides; Refractory Peripheral T-Cell Lymphoma, Not Otherwise Specified; Subcutaneous Panniculitis-Like T-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Enteropathy-Associated T-Cell Lymphoma; Lymphoma, Follicular; Lymphoma, T-Cell; Mycosis Fungoides; Subcutaneous panniculitis-like T-cell lymphoma | interventions — pembrolizumab; 10-propargyl-10-deazaaminopterin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (pralatrexate and pembrolizumab) (Experimental): Patients receive pralatrexate IV over 3-5 minutes on days 1 and 8 and pembrolizumab IV over 30 minutes on day 1. Courses repeat every 21 days for up to 24 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Pembrolizumab; Drug: Pralatrexate

INTERVENTIONS:
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Drug: Pralatrexate — Given IV
  Other Names: 10-propargyl-10-deazaaminopterin; Folotyn; PDX

SUMMARY:
This phase I/II trial studies the side effects and best dose of pralatrexate when given together with pembrolizumab and how well they work in treating patients with peripheral T-cell lymphomas that has come back after a period of improvement or has not responded to treatment. Pralatrexate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving pembrolizumab and pralatrexate may work better in treating patients with peripheral T-cell lymphomas.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the safety and tolerability of a regimen combining pembrolizumab and pralatrexate in patients with relapsed or refractory peripheral T-cell lymphoma (PTCL).

II. Establish the maximum tolerated dose (MTD) and recommended phase II dose (RP2D) of the combined pralatrexate and pembrolizumab regimen.

III. Estimate the overall response rate (ORR) according to the Lugano Classification in patients treated with pembrolizumab plus pralatrexate at the RP2D.

SECONDARY OBJECTIVES:

I. Estimate the complete response (CR) rate according to the Lugano Classification duration of response (DOR), overall survival (OS) and progression-free survival (PFS) in patients treated with pembrolizumab plus pralatrexate.

II. Estimate the ORR and CR rate according to the International Harmonization Project response criteria.

III. Evaluate responses and disease progression according to the Lymphoma Response to Immunomodulatory therapy Criteria (LYRIC).

EXPLORATORY OBJECTIVE:

I. Explore immunologic and genomic biomarkers of response to pembrolizumab plus pralatrexate therapy.

OUTLINE: This is a phase I, dose-escalation study of pralatrexate followed by a phase II study.

Patients receive pralatrexate intravenously (IV) over 3-5 minutes on days 1 and 8 and pembrolizumab IV over 30 minutes on day 1. Courses repeat every 21 days for up to 24 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 and 90 days, every 12 weeks for 1 year, and then every 18 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Documented willingness and ability to sign an informed consent of the participant and/or legally authorized representative.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Patients must have a histologically confirmed diagnosis of mature peripheral T-cell or natural killer (NK)-cell lymphoma according to the World Health Organization (WHO) classification, with hematopathology review at the participating institution. Eligible histologies are:

  * Peripheral T-cell lymphoma, not otherwise specified
  * Anaplastic large cell lymphoma, ALK-negative
  * Anaplastic large cell lymphoma, ALK-positive
  * Angioimmunoblastic T-cell lymphoma
  * Nodal peripheral T-cell lymphoma with TFH phenotype
  * Follicular T-cell lymphoma
  * Indolent T-cell lymphoproliferative disorder of the gastrointestinal (GI) tract
  * Extranodal NK-/T-cell lymphoma
  * Enteropathy-associated T cell lymphoma
  * Monomorphic epitheliotropic intestinal T-cell lymphoma
  * Hepatosplenic T-cell lymphoma
  * Subcutaneous panniculitis-like T-cell lymphoma
  * Transformed mycosis fungoides
* Patients must have failed at least one prior regimen, including:

  * Recurrence of disease after a documented complete response (CR).
  * Progression of disease after a partial response (PR) to the prior regimen.
  * Partial response, stable disease (SD) or progressive disease (PD) at the completion of the prior treatment regimen. If a patient has PR to prior regimen without PD, there must be biopsy-proven** residual disease that is measurable

    * Exception can be granted by the principal investigator (PI) if a biopsy is not feasible and/or safe
* Patient must have measurable disease by computerized tomography (CT) or positron emission tomography (PET) scan, with one or more sites of disease >= 1.5cm in longest dimension.
* Be willing to provide tissue from a fresh core or excisional biopsy of a tumor lesion prior to starting study therapy or from archival tissue of a biopsy that was performed after the most recent systemic therapy. Exception can be granted by the PI if a biopsy is not feasible and/or safe
* Patients must have received one dose of vitamin B12 (1 mg intramuscularly [IM]) within 10 weeks prior to first dose of pralatrexate, and must have begun folic acid supplementation (1 mg orally, once daily) within 10 days of first dose of pralatrexate. Note: If folic acid was not started but methylmalonic acid (MMA) and homocysteine (HCY) levels were checked and are in normal range at screening, the investigator can decide to start study therapy immediately. Vitamin B12 and folic acid supplementation is standard of care for pralatrexate therapy.
* Absolute neutrophil count (ANC) >= 1,000/mm^3. In Phase 2 portion of study, ANC < 1000/mm^3 but >= 500/mm^3 is allowable if patients have demonstrated bone marrow involvement by lymphoma (within 14 days prior to day 1 of protocol therapy).

  * Note: Growth factor is not permitted within 7 days of ANC assessment unless cytopenia is secondary to disease involvement.
* Platelets >= 75,000/mm^3. In Phase 2 portion of study, Platelets < 75,000/mm^3 but >= 25,000/mm^3 is allowable if patients have demonstrated bone marrow involvement by lymphoma (within 14 days prior to day 1 of protocol therapy)

  * Note: Platelet transfusions are not permitted within 7 days of platelet assessment unless cytopenia is secondary to disease involvement.
* Total serum bilirubin =< 1.5 X upper limit of norma (ULN) or =< 3X ULN for Gilbert's disease. Direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN (within 14 days prior to day 1 of protocol therapy).
* Aspartate aminotransferase (AST) =< 2.5 x ULN (within 14 days prior to day 1 of protocol therapy)
* Alanine aminotransferase (ALT) =< 2.5 x ULN (within 14 days prior to day 1 of protocol therapy)
* Creatinine clearance of >= 60 mL/min per the Cockcroft-Gault formula (within 14 days prior to day 1 of protocol therapy). If creatinine clearance (CrCl) is >= 60 mL/min as measured by 24 hour urine collection, this will be allowable.
* If not receiving anticoagulants: International normalized ratio (INR) OR prothrombin (PT) =< 1.5 x ULN (within 14 days prior to day 1 of protocol therapy).

  * If on anticoagulant therapy: PT must be within therapeutic range of intended use of anticoagulants.
* If not receiving anticoagulants: Activated partial thromboplastin time (aPTT) =< 1.5 x ULN (within 14 days prior to day 1 of protocol therapy)

  * If on anticoagulant therapy: aPTT must be within therapeutic range of intended use of anticoagulants.
* Female of childbearing potential: negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication (within 14 days prior to day 1 of protocol therapy). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Woman of childbearing potential (WOCBP): Use two effective methods of contraception (hormonal or barrier method) or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days post last dose of pembrolizumab. WOCBP defined as not being surgically sterilized or have not been free from menses for >1 year.

  * Male: Use two effective methods of contraception (barrier method) or abstain from heterosexual activity with the first dose of study therapy through 120 days post last dose of pembrolizumab.

Exclusion Criteria:

* Patients with adult T-cell leukemia/lymphoma
* Prior allogeneic hematopoietic stem cell transplantation within the last 5 years.
* Prior autologous hematopoietic stem cell transplant within the last 60 days.
* Patients who received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent without having had evidence of objective response.
* Patients who received prior therapy with pralatrexate without having had evidence of objective response.
* Investigational agent or anti-cancer monoclonal antibody (mAb) within 21 days prior to day 1 of therapy or who has not recovered (i.e. =<1 or at baseline) from adverse events due to agents administered more than 21 days earlier.
* Prior chemotherapy, targeted small molecule therapy, or radiation therapy within 14 days prior to day 1 of therapy or who has not recovered (i.e. =< 1 or at baseline) from adverse events due to a previously administered agent. * Note: Subjects with =< grade 2 neuropathy are an exception and may qualify for the study.
* Antineoplastic biologic therapy or major surgery within 21 days of the first dose of trial medication. If subjects received major surgery more than 21 days ago, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Received live vaccine within 30 days prior to day 1 of protocol therapy.
* Systemic steroid therapy or on any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Diagnosis of immunodeficiency.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Congestive heart failure class III/IV according to the New York Heart Association (NYHA) Functional classification.
* Known severe hypersensitivity reaction to pembrolizumab, pralatrexate, leucovorin or any excipients.
* Active autoimmune disease that has required systemic treatment in the past 2 years (replacement therapies for hormone deficiencies are allowed). Hemolytic anemia associated with the lymphoma does not exclude a patient from the study.
* Known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies).
* Known active hepatitis B (e.g., hepatitis B virus surface antigen (HBsAg) reactive) or hepatitis C (e.g., hepatitis C virus ribonucleic acid [HCV RNA] [qualitative] is detected).
* History of tuberculosis (TB) infection (Bacillus tuberculosis).
* Active central nervous system (CNS) involvement by lymphoma, including parenchymal and/or lymphomatous meningitis. Subjects with prior CNS involvement by lymphoma must have a baseline magnetic resonance imaging (MRI) and lumbar puncture at screening that demonstrate no active lymphoma in the CNS.
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Active, uncontrolled infection requires systemic therapy.
* Female: Pregnant or breastfeeding.
* Expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has known psychiatric or substance abuse disorder that would interfere with cooperation with the requirements of the trial.
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures.
* Perspective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2026-02-26 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Alex F Herrera, Principal Investigator — City of Hope Medical Center
Locations (3):
- United States (3):
  - City of Hope Medical Center, Duarte, California
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - University of Nebraska Medical Center, Omaha, Nebraska

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Due to low/slow accrual, this study was permanently closed to accrual after enrolling 13 patients in Phase I, with no accrual in Phase II. Of the 13 patients in Phase I, 7 were at dose level 1 and 6 were at dose level 2.
Groups:
- Phase I - Dose Level 1: Pembrolizumab 200mg + Pralatrexate 20mg/m2: Patients receive pralatrexate 20mg/m2 IV over 3-5 minutes on days 1 and 8 and pembrolizumab 200mg IV over 30 minutes on day 1. Courses repeat every 21 days for up to 24 months in the absence of disease progression or unacceptable toxicity.
- Phase I - Dose Level 2: Pembrolizumab 200mg + Pralatrexate 30mg/m2: Patients receive pralatrexate 30mg/m2 IV over 3-5 minutes on days 1 and 8 and pembrolizumab 200mg IV over 30 minutes on day 1. Courses repeat every 21 days for up to 24 months in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Phase I - Dose Level 1: Pembrolizumab 200mg + Pralatrexate 20mg/m2 | Phase I - Dose Level 2: Pembrolizumab 200mg + Pralatrexate 30mg/m2
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I - Dose Level 1: Pembrolizumab 200mg + Pralatrexate 20mg/m2 | Phase I - Dose Level 2: Pembrolizumab 200mg + Pralatrexate 30mg/m2 | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Continuous [Median (Full Range); unit: years] | 63 [53 to 69] | 68 [49 to 84] | 63 [49 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 6 | 4 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 0 | 5
  Not Hispanic or Latino | 2 | 6 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 6 | 3 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had Dose Limiting Toxicities
Description: Dose limiting toxicities (DLT) were defined as one of the AEs in Protocol Section 5.5 that at least possibly related to study treatment. The DLT observation period was 2 cycles of therapy, from the start of Cycle 1 through the start of Cycle 3. Toxicities were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0).
Time Frame: From the start of Cycle 1 through the start of Cycle 3 (approximately 42 days)
Population: Two patients in dose level 1 and one patient in dose level 2 were not evaluable for DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I - Dose Level 1: Pembrolizumab 200mg + Pralatrexate 20mg/m2 | Phase I - Dose Level 2: Pembrolizumab 200mg + Pralatrexate 30mg/m2
Number analyzed (Participants) | 5 | 5
Participants | 1 | 2

2. Primary Outcome: Number of Participants Who Had Overall Response
Description: Number of participants who had a documented complete response (CR) or partial response (PR) at any time during study treatment. Disease response/progression by PET-CT or CT was evaluated using 2014 Lugano Classification.
Time Frame: Up to 43 months after the initial study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I - Dose Level 1: Pembrolizumab 200mg + Pralatrexate 20mg/m2 | Phase I - Dose Level 2: Pembrolizumab 200mg + Pralatrexate 30mg/m2
Number analyzed (Participants) | 7 | 6
Participants | 2 | 1

3. Secondary Outcome: Number of Participants Who Had Complete Response (CR)
Description: Number of participants who had a documented complete response at any time during study treatment. Disease response/progression by PET-CT or CT was evaluated using 2014 Lugano Classification.
Time Frame: Up to 43 months after the initial study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I - Dose Level 1: Pembrolizumab 200mg + Pralatrexate 20mg/m2 | Phase I - Dose Level 2: Pembrolizumab 200mg + Pralatrexate 30mg/m2
Number analyzed (Participants) | 7 | 6
Participants | 1 | 1

4. Secondary Outcome: Number of Participants With Grade 3 4 5 Adverse Events
Description: Number of Participants who had grade 3 4 5 toxicities at lease possibly related to study treatment. Toxicities were assessed according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Grade refers to the severity of the AE and ranges from 1 to 5 (Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe, Grade 4=Life-threatening, Grade 5=Death).
Time Frame: From the start time of the initial treatment assessed through 8 treatment cycles (21 days per cycle) up to 90 days from last dose (approximately 9 months).
Measure: Number; unit: participants
Arm/Group | Phase I - Dose Level 1: Pembrolizumab 200mg + Pralatrexate 20mg/m2 | Phase I - Dose Level 2: Pembrolizumab 200mg + Pralatrexate 30mg/m2
Number analyzed (Participants) | 7 | 6
participants | 4 | 3

ADVERSE EVENTS:
Time Frame: Adverse Events were assessed through 8 treatment cycles (21 days per cycle) up to 90 days from last dose (approximately 9 months). All-Cause Mortality was monitored/assessed up to 43 months from the start time of the initial treatment.
Arm/Group | Phase I - Dose Level 1: Pembrolizumab 200mg + Pralatrexate 20mg/m2 | Phase I - Dose Level 2: Pembrolizumab 200mg + Pralatrexate 30mg/m2
All-Cause Mortality (participants affected / at risk) | 5/7 | 5/6
Serious Adverse Events (participants affected / at risk) | 2/7 | 3/6
Other Adverse Events (participants affected / at risk) | 7/7 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I - Dose Level 1: Pembrolizumab 200mg + Pralatrexate 20mg/m2 (N=7) | Phase I - Dose Level 2: Pembrolizumab 200mg + Pralatrexate 30mg/m2 (N=6)
CLOSTRIDIOIDES DIFFICILE (Gastrointestinal disorders) | 1 (1) | 0 (0)
DISEASE PROGRESSION (General disorders) | 1 (1) | 1 (2)
FEVER (General disorders) | 1 (1) | 0 (0)
TUMOR FLARE (General disorders) | 0 (0) | 1 (1)
ENCEPHALITIS INFECTION (Infections and infestations) | 1 (1) | 0 (0)
HERPES SIMPLEX REACTIVATION (Infections and infestations) | 0 (0) | 1 (1)
VASCULAR ACCESS COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
LARYNGEAL OBSTRUCTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I - Dose Level 1: Pembrolizumab 200mg + Pralatrexate 20mg/m2 (N=7) | Phase I - Dose Level 2: Pembrolizumab 200mg + Pralatrexate 30mg/m2 (N=6)
ANEMIA (Blood and lymphatic system disorders) | 5 (10) | 1 (1)
EOSINOPHILIA (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
PLATELET COUNT INCREASED (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
SINUS BRADYCARDIA (Cardiac disorders) | 1 (2) | 0 (0)
SINUS TACHYCARDIA (Cardiac disorders) | 3 (10) | 2 (2)
VENTRICULAR ARRHYTHMIA (Cardiac disorders) | 1 (1) | 0 (0)
CATARACT (Eye disorders) | 0 (0) | 1 (1)
PERIORBITAL EDEMA (Eye disorders) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 2 (3) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 3 (3) | 3 (3)
DRY MOUTH (Gastrointestinal disorders) | 1 (1) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 1 (2) | 1 (1)
MUCOSITIS ORAL (Gastrointestinal disorders) | 2 (2) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 2 (3) | 1 (2)
ORAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (2) | 1 (1)
CHILLS (General disorders) | 3 (4) | 0 (0)
DISEASE PROGRESSION (General disorders) | 4 (4) | 2 (2)
EDEMA FACE (General disorders) | 1 (1) | 0 (0)
FACIAL PAIN (General disorders) | 1 (2) | 0 (0)
FATIGUE (General disorders) | 4 (5) | 3 (6)
FEVER (General disorders) | 1 (1) | 1 (2)
GAIT DISTURBANCE (General disorders) | 1 (2) | 0 (0)
GENERALIZED EDEMA (General disorders) | 0 (0) | 1 (1)
MALAISE (General disorders) | 1 (1) | 0 (0)
NECK EDEMA (General disorders) | 1 (1) | 0 (0)
PAIN (General disorders) | 1 (1) | 0 (0)
RASH PUSTULAR (Infections and infestations) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 1 (3) | 0 (0)
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Investigations) | 1 (1) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 2 (4)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 2 (4) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 2 (3) | 1 (2)
BLOOD BILIRUBIN INCREASED (Investigations) | 1 (1) | 0 (0)
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 2 (2) | 1 (1)
CREATININE INCREASED (Investigations) | 0 (0) | 1 (1)
ELECTROCARDIOGRAM QT CORRECTED INTERVAL PROLONGED (Investigations) | 1 (1) | 0 (0)
LYMPHOCYTE COUNT DECREASED (Investigations) | 4 (4) | 1 (1)
NEUTROPHIL COUNT DECREASED (Investigations) | 2 (6) | 1 (4)
PLATELET COUNT DECREASED (Investigations) | 5 (18) | 1 (3)
WEIGHT LOSS (Investigations) | 2 (6) | 0 (0)
WHITE BLOOD CELL DECREASED (Investigations) | 3 (7) | 1 (6)
ANOREXIA (Metabolism and nutrition disorders) | 2 (4) | 3 (3)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPERCALCEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 3 (7) | 2 (2)
HYPERPHOSPHATEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 4 (11) | 1 (1)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 2 (4) | 1 (2)
HYPOKALEMIA (Metabolism and nutrition disorders) | 4 (6) | 1 (1)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 5 (5) | 1 (1)
HYPONATREMIA (Metabolism and nutrition disorders) | 4 (13) | 1 (1)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
OBESITY (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (4) | 1 (1)
HEAD SOFT TISSUE NECROSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCLE CRAMP (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ANAPLASTIC ASTROCYTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
DIZZINESS (Nervous system disorders) | 1 (2) | 1 (1)
DYSARTHRIA (Nervous system disorders) | 1 (1) | 0 (0)
DYSGEUSIA (Nervous system disorders) | 0 (0) | 2 (2)
HEADACHE (Nervous system disorders) | 0 (0) | 1 (1)
HYDROCEPHALUS (Nervous system disorders) | 0 (0) | 1 (1)
HYPERSOMNIA (Nervous system disorders) | 1 (1) | 0 (0)
NEURALGIA (Nervous system disorders) | 1 (1) | 0 (0)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 1 (1) | 0 (0)
ANXIETY (Psychiatric disorders) | 1 (2) | 0 (0)
CONFUSION (Psychiatric disorders) | 1 (4) | 0 (0)
DEPRESSION (Psychiatric disorders) | 1 (1) | 0 (0)
HALLUCINATIONS (Psychiatric disorders) | 0 (0) | 1 (1)
INSOMNIA (Psychiatric disorders) | 0 (0) | 2 (2)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HOARSENESS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
VOICE ALTERATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
BULLOUS DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
HYPERKERATOSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 4 (32) | 1 (5)
HYPOTENSION (Vascular disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-25): https://cdn.clinicaltrials.gov/large-docs/98/NCT03598998/Prot_SAP_000.pdf